CLINICAL TRIAL: NCT06986187
Title: Investigation of Difficult Airway and Difficult Intubation Incidence and Associated Factors in Patients Undergoing Cardiovascular Surgery and a Prediction Model Development
Brief Title: Difficult Airway Incidence in Cardiovascular Surgery and a Prediction Model Development
Acronym: DAPCAP
Status: Recruiting | Type: Observational
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, DILEK YAZICIOGLU, Professor of Anesthesiology, Diskapi Teaching and Research Hospital
Other Study IDs: AEŞH-EK-2025-087
Record Dates: First submitted 2025-05-15; First posted 2025-05-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Difficult Airway Intubation; Difficult Airway; Difficult Intubation; Cardiac Surgery; Cardiac Surgery in Adult Patient
Keywords: difficult intubation; difficult airway; difficult airway prediction; difficult airway prediction model

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A difficult airway is a clinical condition that occurs when one or more of the components of difficult mask ventilation, difficult laryngoscopy, difficult endotracheal intubation, difficult supraglottic airway device (SGA) placement, and inability to intubate-oxygenate are present. Data concerning incidence of difficult airway in patients undergoing cardiovascular surgery is controversial. Unwanted hemodynamic changes that may occur in patients undergoing cardiovascular surgery, combined with hemodynamic changes caused by underlying cardiac pathologies, may also lead to a physiologically difficult airway situation. Since all these interactions, combined with the hemodynamic changes caused by difficult airway interventions, may lead to catastrophic outcomes, it is vital to predict difficult airway in this patient population.

DETAILED DESCRIPTION:
Difficult airway is a clinical condition that occurs when one or more of the components of difficult mask ventilation, difficult laryngoscopy, difficult endotracheal intubation, difficult supraglottic airway device (SGA) placement, and inability to intubate-oxygenate are present.

Different diagnostic criteria for all components of difficult airway and similarly different predictive criteria for the risk of occurrence in a patient have been defined. The LEMON Score, El-Ganzouri Risk Index, and Arne Score, which are evaluated by physical examination of the upper airway structures during the pre-anesthetic examination, and the Cormack-Lehane Classification (CL) used to evaluate the laryngoscopic image during intubation, can be counted among the difficult airway prediction tests.

Difficult airway situations that occur during anesthesia application can be defined by the Han Score for mask ventilation, the Intubation Difficulty Scale (IDS) for endotracheal entubation, the videolaryngoscopic intubation and difficult airway classification (VIDIAC) in patients using videolaryngoscopy, and the difficult SGA placement score.

Previous studies have reported that the incidence of difficult airway is higher in patients undergoing cardiovascular surgery compared to other patient groups. Borde et al. reported the rate of difficult intubation in patients undergoing cardiac surgery as 24%. The rate of difficult laryngoscopy in patients undergoing coronary artery surgery was reported as 10% by Ezri et al. and 7% by Heinrich et al. However, it is seen that the predictive criteria and diagnostic criteria for the components of the difficult airway are used interchangeably and incorrectly in these studies. Therefore, the current information on the incidence of difficult airways in patients undergoing cardiovascular surgery is contradictory and open to debate.

Accurate information on the incidence of difficult airway in this patient population can contribute to anesthesiology education, equipment and personnel planning, and most importantly, patient safety. Unwanted hemodynamic changes that may occur following anesthesia induction in patients undergoing cardiovascular surgery, combined with hemodynamic changes caused by underlying cardiac pathologies, may lead to the emergence of a physiological difficult airway condition. Since all these interactions, when combined with hemodynamic changes caused by difficult airway interventions, may lead to catastrophic outcomes, predicting difficult airway in this patient population is of vital importance.

Despite its clinical importance, to our knowledge, this subject has not yet been investigated in the literature with artificial intelligence algorithms.

The aim of this study is to investigate the incidence of difficult airway and difficult intubation in patients undergoing cardiovascular surgery and the associated factors and to develop a machine learning model that can predict difficult airway using artificial intelligence algorithms.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing cardiovascular surgery
* ASA I-IV physical status
* Over 18 years of age

Exclusion Criteria:

* Known difficult airway
* Head-neck and upper airway pathology
* Patients at risk of aspiration

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery at the Cardiovascular Surgery Department of Etlik City Hospital, Ankara.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Intubation difficulty | 5 minutes after anesthesia induction
  Intubation difficulty is defined with the intubation difficulty scale score and a score greater or equal to 5 is difficult intubation

SECONDARY OUTCOMES:
Dificult mask ventilation | 5 minutes after anesthesia induction
  Difficult mask ventilation is defined by Han scale score, a grade greater or equal to 1 is difficult mask ventilation
Laringeal view score | 5 minutes after anesthesia induction
  Cormack lehanne score will be used , a score greater or equal to 2b is considered predictive of difficult airway
LEMON score | preoperative day
  LEMON score is Look externally Evaluate 3-3-2 rule can 3 fingers fit in the mouth (mouth opening <5 cm) and is the mandible lenght at least 3 fingers from the mentum to the hyoid ( thyromental distance <6 cm) and is the distance from the hyoid to thyroid at least 2 fingers Mallampati class Obstruction (presence of any obstruction) Neck mobility (limited mobility)
  1 point each and >10 points at risk of difficult airway

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Unal, Prof., Principal Investigator — Ankara Etlik City Hospital
Locations (1):
- Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kohse EK, Siebert HK, Sasu PB, Loock K, Dohrmann T, Breitfeld P, Barclay-Steuart A, Stark M, Sehner S, Zollner C, Petzoldt M. A model to predict difficult airway alerts after videolaryngoscopy in adults with anticipated difficult airways - the VIDIAC score. Anaesthesia. 2022 Oct;77(10):1089-1096. doi: 10.1111/anae.15841. Epub 2022 Aug 25. PMID 36006056
- [Background] Cormack RS, Lehane J. Difficult tracheal intubation in obstetrics. Anaesthesia. 1984 Nov;39(11):1105-11. PMID 6507827
- [Background] doi: https://doi.org/10.1097/ALN.0000000000004002